CLINICAL TRIAL: NCT01078935
Title: The Effect of Probiotics on Bowel Disease
Brief Title: The Effect of Probiotics on the Rate of Recovery of Inflammatory Bowel Disease Exacerbation, Endothelial Function, and Markers of Inflammation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Collaborators: Ministry of Health, Israel (Other Government)
Responsible Party: Arnon Blum, The baruch pade medical center, Poriya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Prob-bl.CTIL
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2010-03

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Crohn's disease activity index; CDAI
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: probiotics — Each patient and volunteer will get the study medication for 6 weeks and will be evaluated twice - before enrollment and after 6 weeks of treatment. Routine clinical management will continue - with regular treatment as needed.
Dietary Supplement: placebo — Each patient and volunteer will get the study medication for 6 weeks and will be evaluated twice - before enrollment and after 6 weeks of treatment. Routine clinical management will continue - with regular treatment as needed.

SUMMARY:
Fifty patients will get probiotics (109 bacteria [L. acidophilus, B. bifidum, S. thermophilus, L. rhamnosus, L. casei] in 2 capsules) and half will get placebo (2 capsules that look the same like the probiotic capsules and will contain microcrystalline cellulose, artificial brown color, magnesium strearate, and silica dioxide). The patients and the staff will be blinded to the identity of the study medications.

Each patient and volunteer will get the study medication for 6 weeks and will be evaluated twice - before enrollment and after 6 weeks of treatment. Routine clinical management will continue - with regular treatment as needed.

Each individual will be studied for changes in biochemical inflammatory and immunological markers and changes in flow medicated diameter that will be measured by the brachial artery method (that is evaluating endothelial function). Every patient will be evaluated for his/her ability to produce endothelial progenitor stem cells (EPCs).

ELIGIBILITY:
Inclusion Criteria:

* patients with ulcerative colitis and crohns' disease

Exclusion Criteria:.

* notable caveats are that arteries smaller than 2.5 mm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Truelove and Witts Classification of Ulcerative Colitis | 2 years
Crohn's disease activity index (CDAI) | 2 years